CLINICAL TRIAL: NCT03160105
Title: Evaluation of a Simplified Strategy for the Long-term Management of HIV Infection: a Non-inferiority, Randomized, Controlled, Open-label Clinical Trial
Brief Title: Evaluation of a Simplified Strategy for the Long-term Management of HIV Infection (Simpl'HIV)
Acronym: Simpl'HIV
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Calmy Alexandra (Other)
Responsible Party: Sponsor-Investigator, Calmy Alexandra, Professor, University Hospital, Geneva
Organization: University Hospital, Geneva (Other)
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: CCER 2016-02210
Record Dates: First submitted 2017-05-16; First posted 2017-05-19 (Actual); Last update posted 2019-08-29 (Actual); Status verified 2019-08

CONDITIONS: HIV-1-infection; Antiretroviral Therapy; Maintenance Therapy
MeSH Terms: interventions — Racivir

STUDY DESIGN:
Intervention Model Description: This is a pragmatic multicentre, 2x2 factorial randomized controlled trial with 1:1:1:1 randomization. A sample size of 92 patients in each group will be required to demonstrate non-inferiority with a non-inferiority (NI) margin of 12%.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Continuing cART + Standard monitoring (No Intervention): Patients randomized to this arm will continue their current standard ART regimen (cART) and will continue a standard 3-monthly routine safety biological monitoring (including CD4 cell count, fasting lipids and glucose, renal and hepatic function tests) at their SHCS site.
- Continuing cART + Patient-centered monitoring (Experimental): Patients randomized to this arm will continue their current cART and will have immunological and safety blood examinations performed once per year and at least one options (decentralised venipuncture and blood tests, delivery of ARV drugs by mail and interview by phone or skype call) for weeks 6, 12 and 36
  Interventions: Other: Patient-centered monitoring
- Switch to DTG+FTC + Standard monitoring (Experimental): Patients randomized to this arm will be switched to DTG + FTC dual maintenance therapy and will have immunological and safety blood examinations performed once per year and at least one options (decentralised venipuncture and blood tests, delivery of ARV drugs by mail and interview by phone or skype call) for weeks 6, 12 and 36
  Interventions: Drug: Switch to DTG + FTC
- Switch to DTG+FTC + Patient-centered monitoring (Experimental): Patients randomized to this arm will be switched to DTG + FTC dual maintenance therapy and will have immunological and safety blood examinations performed at screening and at week 48. In addition, patients will be ask to choose at least one of the following alternative options for weeks 6, 12 and 36: decentralised venipuncture and blood tests, delivery of ARV drugs by mail and Assessment and clinical interview by phone or skype call
  Interventions: Drug: Switch to DTG + FTC; Other: Patient-centered monitoring

INTERVENTIONS:
Drug: Switch to DTG + FTC — Switch from standard cART to DTG + FTC dual maintenance therapy.
  Arms: Switch to DTG+FTC + Patient-centered monitoring; Switch to DTG+FTC + Standard monitoring
Other: Patient-centered monitoring — Immunological and safety blood examinations performed only once per year at least one options (decentralised venipuncture and blood tests, delivery of ARV drugs by mail and interview by phone or skype call) for weeks 6, 12 and 36
  Arms: Continuing cART + Patient-centered monitoring; Switch to DTG+FTC + Patient-centered monitoring

SUMMARY:
The purpose of this study is to evaluate whether maintenance antiretroviral therapy could be simplified to DTG + FTC dual therapy and/or patient-centered monitoring once virological suppression is achieved. Using a factorial design, the study aims to assess the efficacy of DTG + FTC dual therapy to maintain virological suppression through 48 weeks of follow-up as well as the costs of a patient-centered ART laboratory monitoring.

DETAILED DESCRIPTION:
This is a pragmatic multicentre, 2x2 factorial randomized controlled trial with 1:1:1:1 randomization to switching to DTG-based maintenance dual therapy in association with FTC or continuation of cART, and to patient-centered monitoring or continuation of standard monitoring.

Patients will be followed during 48 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Informed consent as documented by signature;
2. Documented HIV-1 infection;
3. Enrolled in the Swiss HIV Cohorte Study (SHCS) or receiving care from a medical doctor of the SHCS network;
4. ≥ 18 years of age;
5. HIV-RNA <50 copies/mL at screening and for at least 24 weeks before screening on effective suppressive cART, one blip with less than 200 copies/mL being allowed during this period if followed by at least 2 results < 50 copies/mL.
6. On standard cART at the time of inclusion, i.e.:

   * 2 NRTIs + either 1 NNRTI, 1 boosted PI or 1 INSTI;
   * NRTI-sparing triple ARV regimen (e.g. 1 NRTI + 1 NNRTI + 1 InSTI);
   * Dual therapy with protease inhibitor.

Exclusion Criteria:

1. HIV-2 infection;
2. Previous ART change for unsatisfactory virological response, i.e. slow initial virological suppression, incomplete suppression or rebound. Change of drug or drug class for convenience or toxic effect prevention or management is allowed.

   Note: patients with documented genotype(s) presenting only a M184V mutation remain eligible;
3. Creatinine clearance < 50ml/min;
4. ASAT or ALAT >2.5x upper limit of the norm;
5. Known hypersensitivity, intolerance or allergy to DTG or FTC;
6. Known or suspected non-adherence (defined as <80% adherence, i.e. missed doses > 1x/week) to current treatment in the last 6 months;
7. Concomitant use of drugs that decrease DTG blood concentrations including carbamazepine, oxcarbamazepine, phenytoin, phenobarbital, St John's wort and rifampicin;
8. Women who are pregnant or breast-feeding;
9. a. Presence of any INSTI-resistance. Non-availability of INSTI resistance testing is NOT an exclusion criteria.

   b. Non availability of previous routine resistance test, at least for reverse transcriptase and protease genes.

   Note: Subjects remain eligible in the absence of any previous resistance test only if they are on their first-line antiretroviral regimen;
10. Evidence of acute or chronic hepatitis B virus infection based on results of serology testing.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 186 (Actual)
Dates: Start 2017-05-19 (Actual); Primary Completion 2018-04-18 (Actual); Study Completion 2019-05-20 (Actual)

PRIMARY OUTCOMES:
Efficacy of DTG-based maintenance therapy (< 100 copies/ml) | 48 weeks
  Proportion of patients maintaining HIV-RNA <100 copies/ml throughout 48 weeks
Costs of a patient-centered ART monitoring | 48 weeks
  Direct costs of the two study arms from the health care system perspective at week 48

SECONDARY OUTCOMES:
Efficacy of DTG-based maintenance therapy (<50 copies/ml) | 48 weeks
  Proportion of patients maintaining HIV-RNA <50 copies/ml throughout 48 weeks
Efficacy of DTG-based therapy (<50 copies/ml) by FDA snapshot analysis | 48 weeks
  Proportion of patients with HIV-RNA < 50 cp/ml at week 48
HIV-RNA >100 copies/ml as time to loss of virological response (TLOVR) | 48 weeks
  defined as the first of the two-confirmed HIV-RNA >100 copies/ml (at least two weeks apart)
Change in CD4 cell count | 48 weeks
  from baseline to week 48
Change in HIV-DNA | 48 weeks
  from baseline to week 48
Change in lipidic profile | 48 weeks
  from baseline to week 48
Change in glucose profile | 48 weeks
  from baseline to week 48
Change in Framingham-calculated cardiovascular risk | 48 weeks
  from baseline to week 48
Change in glomerular function rate | 48 weeks
  from baseline to week 48
Proportion of patients with an adverse event | 48 weeks
  throughout week 48
Proportion of patients with a severe adverse event | 48 weeks
  throughout week 48
Proportion of patients with CNS adverse event | 48 weeks
  throughout week 48
Proportion of patients new to DTG with CNS symptoms | 6 weeks
  at 2 and 6 week
PROQOL questionnaire | 48 weeks
  from baseline to weeks 12 and 48
Patient's monitoring satisfaction for pts in the patient-centered monitoring arm | 48 weeks
  from baseline to weeks 24 and 48
Global satisfaction of the monitoring | 48 weeks
  at week 48
Proportion of patients in the patient-centered monitoring arm expressing willingness to change monitoring options | 48 weeks
  Monitoring satisfaction throughout 48 weeks
Patient's treatment satisfaction at week 48 | 48 weeks
  at week 48
ARV treatment in the post study | 48 weeks
  ART decided to be used in the post study period
Study satisfaction | 48 weeks
  at week 48
Cost-effectiveness of study arms | 48 weeks
  at week 48
Change in patient weight | 48 weeks
  from baseline to week 48
Adherence questions | 48 weeks
  Patient adherence to treatment throughout 48 weeks of follow-up
Number of study-related extra clinical visits | 48 weeks
  performed outside trial scheduled throughout 48 weeks

CONTACTS AND LOCATIONS:
Locations (7):
- Switzerland (7):
  - Department of Infectious Diseases and Hospital Epidemiology, University Hospital of Basel, Basel
  - Departement of Infectious Disease, Bern University Hospital, Bern
  - Infectious diseases consultation, University Hospitals of Geneva, Geneva
  - Infectious Diseases Service, Lausanne University Hospital, Lausanne
  - Department of Infectious Diseases, Lugano Regional Hospital, Lugano
  - Division of Infectious Diseases and Hospital Epidemiology, Kantonspital St.Gallen, Sankt Gallen
  - Department of Infectious Diseases and Hospital Epidemiology, University Hospital of Zurich, Zurich

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Marinosci A, Sculier D, Wandeler G, Yerly S, Stoeckle M, Bernasconi E, Braun DL, Vernazza P, Cavassini M, Buzzi M, Metzner KJ, Decosterd L, Gunthard HF, Schmid P, Limacher A, Branca M, Calmy A. Costs and acceptability of simplified monitoring in HIV-suppressed patients switching to dual therapy: the SIMPL'HIV open-label, factorial randomised controlled trial. Swiss Med Wkly. 2024 Apr 15;154:3762. doi: 10.57187/s.3762. PMID 38754068
- [Derived] Sculier D, Wandeler G, Yerly S, Marinosci A, Stoeckle M, Bernasconi E, Braun DL, Vernazza P, Cavassini M, Buzzi M, Metzner KJ, Decosterd LA, Gunthard HF, Schmid P, Limacher A, Egger M, Calmy A; Swiss HIV Cohort Study (SHCS). Efficacy and safety of dolutegravir plus emtricitabine versus standard ART for the maintenance of HIV-1 suppression: 48-week results of the factorial, randomized, non-inferiority SIMPL'HIV trial. PLoS Med. 2020 Nov 10;17(11):e1003421. doi: 10.1371/journal.pmed.1003421. eCollection 2020 Nov. PMID 33170863